CLINICAL TRIAL: NCT03501550
Title: An Open-Label Phase 2a Study Evaluating the Safety and Efficacy of Combination Treatment With 2 Weeks of the Non-Nucleoside Inhibitor CDI 31244 Plus 6 Weeks of Sofosbuvir/Velpatasvir in Subjects With Chronic Hepatitis C Genotype 1 Infection
Brief Title: Study of CDI-31244 in Combination With Sofosbuvir (SOF) and Velpatasvir (VEL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cocrystal Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDI-31244-P2-001
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Chronic Hepatitis C
Keywords: HCV; GT1
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CDI-31244 + SOF/VEL (Experimental): CDI-31244 in combination with SOF/VEL
  Interventions: Drug: CDI-31244; Drug: SOF/VEL

INTERVENTIONS:
Drug: CDI-31244 — investigational drug
  Other Names: CDI-31244 (non-nucleoside inhibitor or NNI)
Drug: SOF/VEL — sofosbuvir and velpatasvir fixed dose combination
  Other Names: Epclusa

SUMMARY:
Open label phase 2a study of two week treatment with CDI-31244 and sofosbuvir and veltapasvir followed by four week treatment of sofosbuvir and velpatasvir in individuals with chronic hepatitis C (HCV) genotype 1 (GT1) infection

DETAILED DESCRIPTION:
The study is open label and has one treatment group. Eligible HCV GT1 subjects will self administer orally 400 mg of CDI-31244 and fixed dose combination of sofosbuvir and velpatasvir for 14 days. After 14 days the subjects will continue the treatment for another 4 weeks on the fixed dose combination sofosbuvir and velpatasvir. The subjects will be followed up until 24 weeks after the last dose of sofosbuvir and velpatasvir to determine if sustained virologic response at 12 (SVR12) and 24 (SVR24) weeks after treatment have been achieved.

ELIGIBILITY:
Key Inclusion Criteria:

Documented chronic HCV GT 1 infection; Serum HCV RNA >1,000 IU/mL during screening; Absence of advanced fibrosis or cirrhosis

Key Exclusion Criteria:

Nursing or pregnant women; Active hepatitis B infection; Human immunodeficiency virus (HIV) infection; History of use of any HCV direct-acting antiviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Chua, MD, Principal Investigator — Institute of Human Virology, University of Maryland, Baltimore
Locations (1):
- Institute of Human Virology University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CDI-31244 + SOF/VEL: 2 wks of CDI-31244 in combination with 6 wks of SOF/VEL
  CDI-31244: investigational drug
  SOF/VEL: sofosbuvir and velpatasvir fixed dose combination
Period: Overall Study
Arm/Group | CDI-31244 + SOF/VEL
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: subjects who received 2 wks of CDI-31244 with 6 wks of SOF and VEL
Groups:
- Subjects: number of subjects in the study
Arm/Group | Subjects
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.08 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
HCV load [Median (Standard Deviation); unit: log10 IU/mL] | 6.59 (0.62)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events
Description: The safety and the tolerability of CDI-31244 in combination with SOF/VEL through number of AEs observed in participants
Time Frame: Day 1 to Day 72
Measure: Count of Participants; unit: Participants
Arm/Group | CDI-31244 + SOF/VEL
Number analyzed (Participants) | 12
Participants | 10

2. Primary Outcome: Number of Participants With Sustained Virologic Response (SVR) 12 Weeks After Treatment
Description: SVR12 is defined as HCV RNA < the lower limit of quantitation (LLOQ) at 12 weeks after treatment
Time Frame: post-treatment Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | CDI-31244 + SOF/VEL
Number analyzed (Participants) | 12
Participants | 8

3. Secondary Outcome: Number of Participants With Sustained Virologic Response (SVR) 24 Weeks After Discontinuation of Therapy
Description: SVR (sustained virologic response) 24 is defined as HCV RNA < the lower limit of quantitation (LLOQ) at 24 weeks after treatment
Time Frame: post-treatment Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | CDI-31244 + SOF/VEL
Number analyzed (Participants) | 12
Participants | 8

ADVERSE EVENTS:
Time Frame: from signing of informed consent to fours weeks after end of treatment (from Study Day 1 to Study Day 72)
Arm/Group | CDI-31244 + SOF/VEL
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDI-31244 + SOF/VEL (N=6)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDI-31244 + SOF/VEL (N=12)
Headache (Nervous system disorders) | 5 (9)
Nausea (Gastrointestinal disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Bunion operation (Surgical and medical procedures) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT03501550/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03501550/SAP_001.pdf